CLINICAL TRIAL: NCT04955119
Title: Fusion Imaging Contrast-enhanced Ultrasound LI-RADS in Patients With High-risk Hepatocellular Carcinoma With Focal Liver Lesions Invisible on Conventional Ultrasound: a Multi-center Prospective Study
Brief Title: Fusion Imaging Contrast-enhanced Ultrasound LI-RADS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: dr.jingxiang003
Record Dates: First submitted 2021-07-03; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fusion imaging contrast-enhanced ultrasound LI-RADS (Experimental): Fusion imaging contrast-enhanced ultrasound will be performed in patients with invisible lesion at conventional ultrasound.
  Drug: SonoVue
  Interventions: Diagnostic Test: Fusion imaging contrast-enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: Fusion imaging contrast-enhanced ultrasound — Fusion imaging contrast-enhanced ultrasound will be performed for patients with invisible lesion at conventional ultrasound.
  Drug: SonoVue

SUMMARY:
CEUS LI-RASD apply to lesion visible at precontrast ultrasound but not the lesion invisible. Fusion imaging can use to invisible lesions at precontrast ultrasound in clinical practice. Thus, our aim is to explore the application value of CEUS LI-RADS in contrast-enhanced fusion imaging for focal liver lesions that are not visible on conventional ultrasound in high-risk patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Patients at risk for HCC(Cirrhosis or Chronic hepatitis B viral infection or Current or prior HCC) Suspicious lesions detected by CECT/MRI but not visible on conventional ultrasound and US-CECT/MRI fusion imaging Patients sign the informed consent.

Exclusion Criteria:

Patients without risk of HCC(With cirrhosis due to congenital hepatic fibrosis or With cirrhosis due to a vascular disorder such as hereditary hemorrhagic telangiectasia, Budd-Chiari syndrome, chronic portal vein occlusion, cardiac congestion, or diffuse nodular regenerative hyperplasia) Patients without a successful registration or lesions can be seen on conventional ultrasound after successful registration Pregnancy or lactation Patients with pretreat lesion Patients don't sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value | 6 months
  The positive predictive value = HCC in LR-5 /all lesions in LR-5

SECONDARY OUTCOMES:
The sensitivity and specificity of CEUS LR-5 | 6 months
  The sensitivity and specificity are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Third Central Hospital, Tianjin, Tianjin Municipality, China